CLINICAL TRIAL: NCT06439745
Title: More Than 50% of the Patients With Clinically Unifocal T1b/Small T2 Node Negative Papillary Thyroid Carcinoma Scheduled for Thyroid Lobectomy May Require Completion Thyroidectomy if the Nodal Status is Evaluated
Brief Title: More Than 50% of Unifocal cN0 T1b/Small T2 Papillary Thyroid Carcinoma May Require Completion Thyroidectomy if Nodal Status is Evaluated
Acronym: cN0PTC
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6584
Record Dates: First submitted 2024-03-07; First posted 2024-06-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-03

CONDITIONS: Papillary Thyroid Cancer; Papillary Carcinoma; Thyroid Cancer; Thyroid Carcinoma; Thyroid Cancer, Papillary; Lymph Node Metastasis
MeSH Terms: conditions — Thyroid Cancer, Papillary; Carcinoma, Papillary; Thyroid Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In absence of nodal metastases or aggressive features, thyroid lobectomy (TL) should be preferred over total thyroidectomy (TT) for small unifocal papillary thyroid carcinoma (PTC). However, occult, despite non-microscopic (>2 mm), nodal metastases may be present in clinically node-negative (cN0) PTCs.

Among 4216 thyroidectomies for malignancy (2014-2023), 110 (2.6%) TL plus ipsilateral central neck dissection (I-CND) were scheduled for unifocal cT1b/small cT2 (<3 cm) cN0 PTCs.

Nodes frozen section examination (FSE) was performed: when positive, completion thyroidectomy (CT) was accomplished during the same procedure. In presence of aggressive pathologic features, CT was suggested within 6 months from index operation.

DETAILED DESCRIPTION:
Papillary thyroid carcinoma (PTC) is the most common type of thyroid cancer. Although its incidence has increased in recent decades, the prognosis is excellent due to the indolent nature of the disease. Despite that, recurrence rate of PTC remains common. Nowadays, the correct extent of thyroidectomy remains controversial. However, several studies demonstrated no significant differences in terms of disease-free survival (DFS) and loco-regional recurrence (LRR) in differentiated thyroid carcinoma (DTC) > 1cm after thyroid lobectomy (TL) vs total thyroidectomy (TT). In absence of preoperative high-risk features (HRFs), the most recent NCCN and ATA guidelines consider unifocal 1-4 cm PTCs eligible for TL. However, many of HRFs are highlighted only after pathological examination: positive nodal status, aggressive tumor subtype, multifocality, microscopic extrathyroidal extension (ETE), positive margin and lymphovascular invasion (LVI).

Recent retrospective series showed that up to 59% of preoperative low risk PCTs were upgraded to higher risk category after pathological examination. Current recommendations could potentially increase the need for re-operation, in terms of completion thyroidectomy (CT) and subsequent administration of RAI in order to reduce the risk of LRR. Among the HRFs, no preoperative clinical parameter is a predictor of nodal disease. However, occult lymph node metastases (LNMs) may be found in 31-62% of patients subjected to prophylactic CND (p-CND). The risk of complications (hypoparathyroidism and laryngeal nerve injury) is the main matter against bilateral p-CND in unifocal node negative PCT. According to a recent systematic review, basing on prevalence of occult central LNM by tumor size, ipsilateral CND (I-CND) may be justified in all PTC patients. Since isolated contralateral metastases are rare, a routine use of frozen section examination (FSE) of I-CND may allow a more accurate staging with a reduction of morbidity. Although p-CND is not usually recommended in patients with clinically unifocal cT1b/T2 node negative PTC, we supposed that the evaluation of LN status through FSE of I-CND may significantly contribute to risk stratification and consequently to modulate the extension of surgical treatment.

In this retrospective study we aim to evaluate the result of this strategy to intraoperatively identify patients who may benefit from TT with bilateral CND (B-CND), reducing the need of second step CT and, theoretically, the risk of LRR.

Among 4176 patients who underwent thyroidectomy for malignancy between September 2014 and September 2023 at Fondazione Policlinico Universitario A. Gemelli - Rome, we identified 110 patients scheduled for TL plus I-CND for clinically intrathyroidal unifocal cT1b/small cT2 node negative PTC. Every patient was informed of the risks and benefits of TL and TT, based on available guidelines.

Inclusion criteria were: age>18; classic papillary carcinoma and variants; clinically unifocal and intrathyroidal PTC; clinical tumor size >1 cm and ≤3 cm; no clinical evidence of LN involvement.

Exclusion criteria were: age < 18 years; prior head or neck irradiation; family history of thyroid carcinoma; clinical evidence of multifocality, extrathyroidal extension or LN metastases; follow-up < 6 months.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* classic papillary carcinoma and variants
* clinically unifocal and intrathyroidal PTC
* clinical tumor size >1 cm and ≤3 cm
* no clinical evidence of LN involvement

Exclusion Criteria:

* age < 18
* prior head or neck irradiation
* family history of thyroid carcinoma
* clinical evidence of multifocality
* extrathyroidal extension or LN metastases
* follow-up < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical treatment of papillary thyroid carcinoma at the Surgical Division of Endocrine and Metabolic Surgery of Fondazione Policlinico Universitario A. Gemelli IRCCS between September 2014 and September 2023.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
evaluation of patients requiring total thyroidectomy | September 2014-September 2023
  Evaluation of histopathologic risk factors in patients with papillary thyroid carcinoma, consisting of rate of nodal metastases, aggressive variants, lympho-angioinvasion, extranodal extension, multifocalty, positive resection status, in order to tailor surgical strategy (completion thyroidectomy)

SECONDARY OUTCOMES:
evaluation of disease recurrence | September 2014-September 2023
  Evaluation of the rate of disease recurrence among the patients' cohort

IPD SHARING:
Plan to Share IPD: Undecided